CLINICAL TRIAL: NCT07321327
Title: Implementation Strategies for Caregiver and Teacher Use of Behavioral Interventions: Aim 2
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 25-023858
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Attention Deficit Hyperactivity Disorder Symptoms
Keywords: Attention Deficit Hyperactivity Disorder Positive Behavior Management; Inattentive; Hyperactive; Impulsive
MeSH Terms: conditions — Spasm; Impulsive Behavior | interventions — Caregivers

STUDY DESIGN:
Intervention Model Description: Participating teachers, and the students and students' caregivers nested within their classroom, are randomized to one of two conditions: implementation strategy resource package for teacher and caregiver, or implementation strategy resource package for teacher only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Teachers in this group will receive an implementation support package and receive support in using it within their classroom management practice. Also within the intervention group (experimental), will be up to 2 students nested in the classroom and their caregivers. Caregivers in this group will receive an implementation support package and receive support in using it.
  Interventions: Behavioral: Positive Behavior Management Toolkit for Caregivers; Behavioral: Positive Behavioral Management Toolkit for Teachers
- Control Group (Active Comparator): Teachers in this group will receive an implementation support package and receive support in using it within their classroom management practice. Also within the control group (active comparator) will be up to 2 students nested in the classroom and their caregivers. Caregivers in this group will not receive the implementation resource package.
  Interventions: Behavioral: Positive Behavioral Management Toolkit for Teachers

INTERVENTIONS:
Behavioral: Positive Behavior Management Toolkit for Caregivers — The Positive Behavior Management Toolkit for Caregivers, or the implementation strategy resource package for caregivers, is a set of resources provided that aims to support their use of evidence-based behavior management practices and home-school communication strategies.
  Other Names: Implementation Strategy Resource Package for Caregivers; Supporting School Success - Caregiver Version (SSS-C)
  Arms: Intervention Group
Behavioral: Positive Behavioral Management Toolkit for Teachers — The Positive Behavior Management Toolkit for Teachers, or the implementation strategy resource package for teachers, is a set of resources provided that aims to support their use of evidence-based behavior management practices and home-school communication strategies.
  Other Names: Implementation Strategy Resource Package for Teachers; Supporting School Success - Teacher Version (SSS-T)

SUMMARY:
The purpose of this study is to pilot test for feasibility and initial promise an implementation strategy resource package that aims to support caregivers in using behavioral interventions for children with hyperactive, inattentive, or impulsive behaviors, when provided as an adjunct to a resource package for teachers. Participating children will be randomized at the classroom level to one of two conditions: a) their teacher and caregiver receive the resource package, or b) only their teacher receive the resource package. The research team will examine teacher and caregiver implementation outcomes and mental health outcomes for enrolled children.

DETAILED DESCRIPTION:
Evidence-based interventions for children with or at-risk for Attention Deficit Hyperactivity Disorder (ADHD) include antecedent- and consequence- based behavioral interventions in both the classroom and home settings as well as effective home-school communication approaches. Schools are a promising setting in which to provide early intervention for mental health challenges and to increase access to mental health care. Furthermore, stronger integration between home- and school- based interventions has the potential to meaningfully improve child outcomes. However, there are substantial implementation challenges to caregivers' use of these evidence-based interventions. The purpose of this study is to pilot test for feasibility and initial promise an implementation strategy resource package that aims to support caregivers in using behavioral interventions for children with hyperactive, inattentive, or impulsive behaviors, when provided as an adjunct to a resource package for teachers. Participating children will be randomized at the classroom level to one of two conditions: a) both teacher and caregiver receive the resource package, or b) only the teacher receive the resource package. The research team will examine teacher and caregiver implementation outcomes and mental health outcomes for enrolled children.

ELIGIBILITY:
Teacher Inclusion criteria

* A K-5 teacher at a participating school
* Informed consent

Child Inclusion Criteria

* Is in a K-5 (ages 4-13 years) class of a participating teacher
* Nominated for participation by the participating teacher
* Identified by their participating teacher as displaying functional impairment from ADHD symptoms, as measured by a score of a 3 or greater on the modified version of the Impairment Rating Scale.
* Informed consent and assent if appropriate

Child Exclusion Criteria

* Special education classification of 'intellectual disability'
* Presents as in acute risk of harm to self or others, such that participation in the study is clinically inappropriate because the child warrants more intensive intervention
* Students from families in which there is not a caregiver who speaks English will be excluded because the focus of this study is developing an English-language version of the resource package

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-03 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure - Caregiver Report | Endpoint (i.e., at least 8 weeks from resource package receipt)
  Caregiver-reported total score on the Feasibility of Intervention Measure (FIM), which consists of 4 items on a 5-point Likert scale (from 1 = Completely Disagree to 5 = Completely Agree). The total score is the average of the 4 item scores (possible range: 1 through 5, where 5 is the best possible outcome).
Feasibility of Intervention Measure - Teacher Report | Endpoint (i.e., at least 8 weeks from resource package receipt)
  Teacher-reported total score on the Feasibility of Intervention Measure (FIM), which consists of 4 items on a 5-point Likert scale (from 1 = Completely Disagree to 5 = Completely Agree). The total score is the average of the 4 item scores (possible range: 1 through 5, where 5 is the best possible outcome).
Acceptability of Intervention Measure - Caregiver Report | Endpoint (i.e., at least 8 weeks from resource package receipt)
  Caregiver-reported total score on the Acceptability of Intervention Measure (AIM), which consists of 4 items on a 5-point Likert scale (from 1 = Completely Disagree to 5 = Completely Agree). The total score is the average of the 4 item scores (possible range: 1 through 5, where 5 is the best possible outcome).
Acceptability of Intervention Measure - Teacher Report | Endpoint (i.e., at least 8 weeks from resource package receipt)
  Teacher-reported total score on the Acceptability of Intervention Measure (AIM), which consists of 4 items on a 5-point Likert scale (from 1 = Completely Disagree to 5 = Completely Agree). The total score is the average of the 4 item scores (possible range: 1 through 5, where 5 is the best possible outcome).
Intervention Appropriateness Measure - Caregiver Report | Endpoint (i.e., at least 8 weeks from resource package receipt)
  Caregiver-reported total score on the Intervention Appropriateness Measure (IAM), which consists of 4 items on a 5-point Likert scale (from 1 = Completely Disagree to 5 = Completely Agree). The total score is the average of the 4 item scores (possible range: 1 through 5, where 5 is the best possible outcome).
Intervention Appropriateness Measure - Teacher Report | Endpoint (i.e., at least 8 weeks from resource package receipt)
  Teacher-reported total score on the Intervention Appropriateness Measure (IAM), which consists of 4 items on a 5-point Likert scale (from 1 = Completely Disagree to 5 = Completely Agree). The total score is the average of the 4 item scores (possible range: 1 through 5, where 5 is the best possible outcome).
Change in teacher-report child performance | Baseline, endpoint (i.e., at least 8 weeks from resource package receipt)
  Teacher-reported performance items on the National Institute for Children's Health Quality Vanderbilt Scale - Teacher Version; These 8 items are rated on a 5-point scale (from 1 = Excellent to 5 = Problematic). The total score is the average of the 8 item scores (possible range 1 through 5, where 1 is the best possible outcome).
Change in caregiver-report child performance | Baseline, endpoint (i.e., at least 8 weeks from resource package receipt)
  Caregiver-reported performance items on the National Institute for Children's Health Quality Vanderbilt Scale - Parent Version; These 7 items are rated on a 5-point scale (from 1 = Excellent to 5 = Problematic). The total score is the average of the 7 item scores (possible range 1 through 5, where 1 is the best possible outcome).
Change in teacher-reported parent-teacher relationship | Baseline, endpoint (i.e., at least 8 weeks from resource package receipt)
  Teacher-reported items on a 5-item subscale from the Parent-Teacher Involvement Questionnaire. These 5 items are rated on a 5-point scale (from 0 to 4). The total score is the average of the 5 item scores (possible range 0 to 4, where 4 is the best possible outcome).
Change in caregiver-reported parent-teacher relationship | Baseline, endpoint (i.e., at least 8 weeks from resource package receipt)
  Caregiver-reported items on a 6-item subscale from the Parent-Teacher Involvement Questionnaire. These 6 items are rated on a 5-point scale (from 0 = "not at all" to 4 = "a great dael"). The total score is the average of the 6 item scores (possible range 0 to 4, where 4 is the best possible outcome).
Change in academic productivity | Baseline, endpoint (i.e., at least 8 weeks from resource package receipt)
  Teacher-reported Academic Productivity subscale score of the Academic Performance Rating Scale (APRS). The Academic Productivity subscale includes 12 items, each rated on a 5-point Likert scale from 1 to 5. Four items are reverse scored, and the total score is computed as the average of the 12 items (possible range: 1 through 5, where 5 is the best possible outcome).

SECONDARY OUTCOMES:
Change in Caregiver-reported ADHD symptoms | Baseline, endpoint (i.e., at least 8 weeks from resource package receipt)
  Caregiver-reported inattention and hyperactivity/impulsivity symptoms scores on the National Institute for Children's Health Quality Vanderbilt Scale - Parent Version, which consists of 18 items, rated on 4-point scales (from 0 = Never to 3 = Very Often). The total score is calculated as the average of the of the 18 item scores (possible range 0 through 3, where 0 is the best possible outcome).
Change in Teacher-reported ADHD symptoms | Baseline, endpoint (i.e., at least 8 weeks from resource package receipt)
  Teacher-reported inattention and hyperactivity/impulsivity symptoms scores on the National Institute for Children's Health Quality Vanderbilt Scale - Teacher Version, which consists of 18 items, rated on 4-point scales (from 0 = Never to 3 = Very Often). The total score is calculated as the average of the of the 18 item scores (possible range 0 through 3, where 0 is the best possible outcome).
Change in Student-Teacher Relationship | Baseline, endpoint (i.e., at least 8 weeks from resource package receipt)
  Teacher-reported total score on the Student-Teacher Relationship Scale - Short form, which consists of 15 items, rated on a 5-point scale (from 1 = Definitely does not apply to 5 = Definitely applies). Eight items are reverse scored and then the total score is computed as the average of the 15 item scores (possible range: 1 through 5, where 5 is the best possible outcome).
Change in academic success | Baseline, endpoint (i.e., at least 8 weeks from resource package receipt)
  Teacher-reported Academic Success subscale score of the Academic Performance rating Scale (APRS). The Academic Success subscale includes 7 items, each rated on a 5-point Likert scale from 1 to 5. One item is reverse scored, and the total score is computed as the average of the 7 items (possible range: 1 through 5, where 5 is the best possible outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided